CLINICAL TRIAL: NCT06071299
Title: Impact of Family-Centered Care for Intimate Partner Violence (IPV)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2000035185; 1K23HD107178-01A1 (NIH)
Record Dates: First submitted 2023-09-29; First posted 2023-10-06 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Intimate Partner Violence

STUDY DESIGN:
Intervention Model Description: An anticipated 100 caregivers and 100-150 children of these caregivers, and 85 professionals. Participants will be randomized (1:1) child-caregiver dyads who are reported to the New Haven, Milford and Hartford child protective services (CPS) offices after identified exposure to IPV to either the FCC model or usual child-focused care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FCC model (Experimental): Participants will receive family-focused care.
  Interventions: Behavioral: FCC
- CCC model (Active Comparator): Participants will receive the usual child-focused care.
  Interventions: Behavioral: CCC

INTERVENTIONS:
Behavioral: FCC — Children evaluated for abusive injuries. Caregiver offered meeting with IPV advocate during visit (survivor-centered care, immediate access to services; continued engagement with advocate for ongoing needs). Referral to Child-Study center for trauma follow up. Connection to pediatrician. Use of motivational interviewing to address IPV.
  Arms: FCC model
Behavioral: CCC — Children evaluated for abusive injuries. Medical provider offers IPV resources to caregiver. Referral to Child-Study center for trauma follow up. Connection to pediatrician. Use of motivational interviewing to address IPV.
  Arms: CCC model

SUMMARY:
The purpose of the study will be to determine how participation in Family-Centered Care (FCC) compared to Child-centered care (CCC) will affect caregiver engagement in IPV-based community services, caregiver perceptions of empowerment and survivor-defined practice, and clinical outcomes for children exposed to IPV.

DETAILED DESCRIPTION:
The study population includes victims of intimate partner violence whose children < 5-years old have been referred to Child Protective Services due to exposure to IPV and who have agreed to a medical evaluation for the child(ren) in the child advocacy center or the SCAN clinic and don't already have a connection to an IPV advocate. The study population will include adults who are primarily English or Spanish Language preferring. For professionals, the target audience will be local CPS investigators in the New Haven and Hartford CPS office, IPV advocates at the New Haven Umbrella Center for Intimate Partner Violence Services and The Hartford Interval House and child abuse pediatricians at Yale University School of Medicine and at the Connecticut Childrens Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* Have a child < 5-years-old who been reported to Child Protectives Services for IPV exposure
* Parent > 18 years old who has agreed to a medical evaluation for the child at the child advocacy center
* Does not already have a connection to an IPV advocate
* Able to speak English or Spanish fluently
* Not a ward of department of children and families

Exclusion Criteria:

* Ward of the state
* Language preference other than English or Spanish

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of caregivers with follow-up visits with an IPV advocate | up to 3 months post visit 1
  Percentage of caregivers who have at least one follow-up visit with an IPV advocate by 3 months after the initial visit by self-report.

SECONDARY OUTCOMES:
Percentage of evaluated children who complete a skeletal survey | up to 4 weeks post visit 1
  Percentage of evaluated children <1 yr who complete a skeletal survey up to 4 weeks after the initial visit.
Perceptions of survivor-defined practice using the Survivor Defined Practice Scale (SDPS) | up to 4 weeks post visit 1
  The SDPS is a nine-item measure that assesses intimate partner violence survivors' perception of the degree to which their advocates help them achieve goals they set for themselves, facilitate a spirit of partnership, and show sensitivity to their individual needs and styles. Items are scored on a scale of 1-4 (strongly disagree to strongly agree). Total score range of 9-36. Higher scores indicate a better perception of advocates help.
Perceptions of safety-related empowerment using the Measure of Victim Empowerment Related to Safety (MOVERS) scale. | up to 4 weeks post visit 1
  MOVERS is a 13-item scale that measures survivor empowerment within the domain of safety. MOVERS is composed of three subscales that assess distinct domains of safety related empowerment: Internal Tools, Expectation of Support, and Trade-offs. Participants respond to each item using a five-point Likert scale (from "never true" to "always true") with the Trade-offs subscale being reversed scored. Scores on each subscale are summed to produce total scores. Higher scores indicate an increase in safety related empowerment.
Frequency of IPV-related episodes assessed using the Psychological Maltreatment of Women Inventory (PMWI)- Short form | up to 1 year post visit 1, until child is 2 years of age
  The PMWI is a 14 item questionnaire that assesses psychological maltreatment. Response options on a 5-point Likert scale, ranging from never (1) to very often (5), for the last 6 months. Total score range from 14-70 with higher scores indicating more psychologically abusive experiences.
Frequency of IPV-related episodes assessed using the Conflict Tactic Scale 2 (CTS2) for partner's behaviors | up to 1 year post visit 1, until child is 2 years of age
  The physical assault portion of the CTS2 is a 12 item questionnaire assessing chronicity and prevalence of IPV. Each item is scored on an 7-point Likert scale, ranging from 0 (never) to 6 (>20 times). Only items referring to the partner's behaviors will be included. Total scores range from 0-300 (for chronicity) and 0-12 (for prevalence) with higher scores denoting increased frequency of intimate partner violence.
Number of reports to Child Protective Services (CPS) for IPV | up to 1 year post visit 1
  Number of reports called in to Child Protective Services (CPS) for IPV that identified child as a victim within one year of visit.

CONTACTS AND LOCATIONS:
Overall Officials: Gunjan Tiyyagura, MD, MHS, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - SCAN Clinic, Hartford, Connecticut
  - The South Central Child Advocacy Center, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No